CLINICAL TRIAL: NCT00772980
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Evaluation of the Efficacy, Safety and Tolerability of Neramexane in Patients With Subjective Tinnitus
Brief Title: Efficacy, Safety and Tolerability of Neramexane in Comparison to Placebo in Patients With Subjective Tinnitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. Irena Pulte, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRZ 92579/TI/3002; EudraCT Number 2008-000639-16
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Subjective Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug: Neramexa mesylate Double-blind treatment period of 17 weeks up to 75 mg Neramexane mesylate per day
  Interventions: Drug: Neramexane mesylate
- 2 (Placebo Comparator): Drug: Placebo Double-blind treatment period of 17 weeks placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neramexane mesylate — Double-blind treatment period of 17 weeks up to 75 mg Neramexane mesylate per day, 12 weeks follow-up.
  Arms: 1
Drug: Placebo — Double-blind treatment period of 17 weeks placebo, 12 weeks follow-up.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of neramexane mesylate in the treatment of subjective tinnitus in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 75 years with a clinical diagnosis of first onset, persistent (i.e. tinnitus sghould never be absent for >24 hours in a row), subjective, uni-or bilateral tinntius present for at least 3 months but not more than 12 months.

Exclusion Criteria:

* Clinical diagnosis of intermittent or pulsatile tinnitus
* Patients who have tinnitus as a concomitant symptom of an otological/neurological disease(such as otitis media, Meniére´s disease, otosclerosis, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
TBF-12 (Tinnitus-Beeinträchtigungs-Fragebogen-12 "Tinnitus Handycap Inventory-12") total score change from baseline to end of treatment | Screening, Baseline, week 5, 13, 17

SECONDARY OUTCOMES:
TBF-12 factorial scores, individual respond rate, Tinnitus Rating Scale, Sleep Questionnaire, Qualitiy Of Life, population pharmacokinetics, optional pharmacogenetics | 29 weeks
safety parameters | 29 weeks

CONTACTS AND LOCATIONS:
Locations (55):
- Belgium (8):
  - AZ Sint Lucas, ENT department, Assebroek-Brugge
  - University Hospital Brussels, ENT department, Brussels
  - Clinique Universitaire Saint-Luc, Brussels
  - Dr. Henri HABERMAN, Brussels
  - AZ Sint Lucas, ENT department, Ghent
  - Centre hospitalier de jolimont, La Louvière
  - University Hospital Leuven, ENT Department, Leuven
  - CHU Liege Service ORL, Liège
- Czechia (10):
  - Medico, Chodov, Prague
  - Prof. MUDr. Ivo Šlapák, CSc, Brno
  - Teaching University Hospital, ORL klinika, Brno
  - Nemocnice Havlíčkův Brod, Havlíčkův Brod
  - ORL - Otorynolaryngologické oddělení, Jihlava
  - ORL oddělení, Karlovarská krajská nemocncie a.s., Karlovy Vary
  - Oblastní nemocnice Kladno a.s., Kladno
  - Pro-audio,s.r.o.-private ENT clinic, Mladá Boleslav
  - ORL oddělení, Všeobecná Fakultní Nemocnice v Praze, Prague
  - ORL oddělení , Karlovarská krajská nemocnice a. s., Sokolov
- France (10):
  - Dr. Ebbo, Issy-les-Moulineaux
  - Dr. Sarfati, La Seyne-sur-Mer
  - Centre Hospitalier de Bretagne Sud Service, Lorient
  - Hopital Edouard Herriot, Lyon
  - BONFILS, Paris
  - OHRESSER, Paris
  - Hopital Nord, Saint-Etienne
  - FRAYSSE, Toulouse
  - Service ORL CHU, Tours
  - Hopital Paul BROUSSE Polyclinique, Villejuif
- Netherlands (7):
  - Andromed Breda, Breda
  - Andromed Leiden, Leiderdorp
  - Rijnland Ziekenhuis, ENT department, Leiderdorp
  - Adromed Nijmegen, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer
- Poland (14):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej Prywatne Centrum Medyczne PROMEDIS, Gdansk
  - Szpital Miejski im. J.Brudzinskiego, Gdynia
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - NZOZ Specjalistyczne Centrum Medyczne Nowomed, Krakow
  - Specjalistyczny Gabinet Otolaryngologiczny Dr Anna Otto- Markiewicz, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej PROMED, Krakow
  - Szpital Specjalistyczny im. Stefana Zeromskiego, SP ZOZ w Krakowie, Oddzial Otolaryngologii, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Instytut Medycyny Pracy im. Prof. Dr med. Jerzego Nofera w Lodzi, Lodz
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynała Wyszynskiego Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Instytut Fizjologii i Patologii Sluchu, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
- South Africa (6):
  - Louis Leipoldt Mediclinic, Bellville
  - Lakeview Hospital, Benoni
  - Dr. A. Viljoen, Pretoria
  - GCT Eastmed Clinical Trial centre, Pretoria
  - Constantiaberg Medi Clinic, Western Cape
  - Dr. J. Steer, Wynberg